CLINICAL TRIAL: NCT06856044
Title: Etude Prospective Exploratoire Pilote de sécurité, d'Une Chirurgie Emportant le mésentère Chez Les Patients Porteurs d'Une Maladie de Crohn Avec Atteinte iléo-colique Sous biothérapie
Brief Title: Safety of Mesentery-embedding Surgery in Patients With Ileocolic Crohn's Disease on Biotherapy
Acronym: RIC-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2023-2/MB-01
Record Dates: First submitted 2024-11-29; First posted 2025-03-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with Crohn Disease (Experimental)
  Interventions: Procedure: ileocolic resection with extended mesenteric resection

INTERVENTIONS:
Procedure: ileocolic resection with extended mesenteric resection — The resection limits will be in healthy mesenteric areas. The restoration of continuity in one stage should be preferred. The choice of laparoscopy versus laparotomy is at the surgeon's discretion.

SUMMARY:
60% of patients with Crohn's disease will undergo surgery during their lifetime and without recurrence prevention treatment, 80% of patients will have an endoscopic recurrence within 1 year of surgery. This procedure is performed as close as possible to the gastrointestinal tract, but remaining mesenteric disease is a risk factor for recurrence. Mesentery resection has encouraging results on recurrence requiring reoperation, with a reduction of over 30% in recurrences compared with the standard technique. The study authors wish to evaluate the safety of ileocolic resection surgery involving the mesentery in patients with Crohn's disease treated with biotherapy.

The study hypothesis is that mesentery surgery is no more risky than conventional (gold standard) surgery, and reduces the 6-month endoscopic recurrence rate in patients with ileocolic Crohn's disease on biotherapy requiring ileocolic resection.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient with histologically proven Crohn's disease
* Patient who has undergone ileocolic resection and whose disease site is accessible to endoscopic follow-up (first or repeat operation)
* Patient on anti-TNF α: infliximab or adalimumab (ECCO 2014 recommendation), vedolizumab, ustkinumab, or other biotherapy (e.g. risankizumab)
* Patient able to understand, write and read French

Exclusion Criteria:

* The patient is participating in an interventional study
* The patient is under safeguard of justice or state guardianship
* Medical treatment other than biotherapies including anti-TNF α (infliximab or adalimumab), vedolizumab, ustkinumab, risankinumab
* Contraindication to surgery, such as major cardiovascular comorbidities
* Pregnant, breast-feeding or parturient women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Post-surgical complication rate | 30 days after surgery
  Percentage, graded according to the Clavien-Dindo Classification

SECONDARY OUTCOMES:
Postoperative endoscopic recurrence | 6 months
  Yes/No according to Rutgeerts classification (i0-i4), using a cut-off score ≥ i2
Surgical time of the ileocolic resection technique | End of surgery
  Minutes
Intraoperative bleeding | End of surgery
  If yes, volume (ml)
Length of hospital stay | End of hospitalization (max 1 month)
  Days
Presence of intra- and post-operative complications | Immediately following surgery
  Yes/no
Number of intra- and post-operative complications | Immediately following surgery
  Number
Time until resumption of transit following surgery | Following surgery (maximum 5 days)
  Number of days between surgery and resumption of transit
Time until resumption of eating | Following surgery (average 1 day)
  Number of days between surgery and resumption of eating
Presence of myenteric plexitis with at least one inflammatory cell at proximal ileal resection margin | Immediately following surgery
  Classed as: Absent; 1-3 inflammatory cells; 4-9; or 10+
Number of lymph nodes in the histological specimen | Immediately following surgery
  Number
Resection not in healthy margin | Immediately following surgery
  (Yes/No)
Length of resected digestive tract | Immediately following surgery
  Centimeters
Area of mesentery removed | Immediately following surgery
  Square centimeters
C-reactive protein level | Day before surgery
C-reactive protein level | Day 2
C-reactive protein level | Day 4
C-reactive protein level | Month 1
C-reactive protein level | Month 6
Albuminemia | Day before surgery
Hemoglobinemia | Day before surgery
Hemoglobinemia | Day 2
Hemoglobinemia | Day 4
White blood cells | Day before surgery
White blood cells | Day 2
White blood cells | Day 4
Fecal calprotectin | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Martin BERTRAND, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - CHU de Montpellier Hôpital St Eloi, Montpellier
  - CHU de Nîmes, Nîmes